CLINICAL TRIAL: NCT00494871
Title: Evaluation of the Efficacy and Safety of Rivaroxaban (BAY59-7939) for the Prevention of Stroke and Non-central Nervous System Systemic Embolism in Subjects With Non-valvular Atrial Fibrillation
Brief Title: Efficacy and Safety of Rivaroxaban for the Prevention of Stroke in Subjects With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen R&D, L.L.C. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12620
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
Keywords: BAY59-7939; Rivaroxaban; Non-Valvular Atrial Fibrillation; Japanese Patients; Phase III; 12620
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Participants received once daily (OD) a rivaroxaban 15 mg tablet and a warfarin placebo tablet during the double-blind treatment period
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Warfarin placebo
- Warfarin (Active Comparator): Participants received OD a warfarin potassium tablet and a rivaroxaban placebo tablet during the double-blind treatment period
  Interventions: Drug: Warfarin; Drug: Rivaroxaban placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Participants orally administered rivaroxaban 15 mg OD (CrCL [creatinine clearance] >= 50 mL/min) or 10 mg OD (CrCL 30-49 mL/min)
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Warfarin — Participants orally administered a warfarin potassium tablet (INR [international normalized ratio] target was 1.6-2.6 for patients >70 years and 2.0-3.0 for patients <70 years)
  Arms: Warfarin
Drug: Rivaroxaban placebo — Participants orally administered a rivaroxaban placebo tablet
  Arms: Warfarin
Drug: Warfarin placebo — Participants orally administered a warfarin placebo tablet (adjusted based upon sham INR values)
  Arms: Rivaroxaban (Xarelto, BAY59-7939)

SUMMARY:
This is a clinical study evaluating the efficacy and safety of rivaroxaban for stroke prevention in patients with atrial fibrillation (originally described in Japanese).

DETAILED DESCRIPTION:
Within the US 'Johnson & Johnson Pharmaceutical Research & Development, L.L.C.' is sponsor.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Japanese male or female
* Non- valvular atrial fibrillation documented by ECG
* Patients with a risk of stroke and non-CNS systemic embolism

Exclusion Criteria:

* Significant mitral stenosis
* Patients in whom anticoagulants are contraindicated

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (116):
- Japan (116):
  - Kasugai, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Goshogawara, Aomori
  - Hirosaki, Aomori
  - Asahi, Chiba
  - Funabashi, Chiba
  - Imba, Chiba
  - Matsudo, Chiba
  - Yotsukaidō, Chiba
  - Imabari, Ehime
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Saijō, Ehime
  - Tōon, Ehime
  - Fukui-shi, Fukui
  - Chikushi-gun, Fukuoka
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Ogōri, Fukuoka
  - Yame, Fukuoka
  - Kōriyama, Fukushima
  - Gifu, Gifu
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Mebashi, Gunma
  - Ōtake, Hiroshima
  - Asahikawa, Hokkaido
  - Chitose, Hokkaido
  - Hakodate, Hokkaido
  - Muroran, Hokkaido
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Sunagawa, Hokkaido
  - Tomakomai, Hokkaido
  - Kobe, Hyōgo
  - Higashiibaraki, Ibaraki
  - Hitachi, Ibaraki
  - Jōsō, Ibaraki
  - Kasama, Ibaraki
  - Moriya, Ibaraki
  - Namegata, Ibaraki
  - Toride, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Nomi, Ishikawa-ken
  - Hanamaki, Iwate
  - Morioka, Iwate
  - Marugame, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Izumi, Kagoshima-ken
  - Kagoshima, Kagoshima-ken
  - Atsugi, Kanagawa
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Nangoku, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Uji, Kyoto
  - Kuwana, Mie-ken
  - Sendai, Miyagi
  - Komoro, Nagano
  - Matsumoto, Nagano
  - Suwa, Nagano
  - Nagasaki, Nagasaki
  - Jōetsu, Niigata
  - Nagaoka, Niigata
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Yufu, Oita Prefecture
  - Kasaoka, Okayama-ken
  - Okayama, Okayama-ken
  - Okinawa, Okinawa
  - Shimajiri, Okinawa
  - Daitō, Osaka
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Kawachi-Nagano, Osaka
  - Kishiwada, Osaka
  - Osaka, Osaka
  - Takatsuki, Osaka
  - Toyonaka, Osaka
  - Yao, Osaka
  - Hanyū, Saitama
  - Kasukage, Saitama
  - Kitamoto, Saitama
  - Tokorozawa, Saitama
  - Wako, Saitama
  - Kusatsu, Shiga
  - Fujinomiya, Shizuoka
  - Fukuroi, Shizuoka
  - Hamamatsu, Shizuoka
  - Iwata, Shizuoka
  - Shimada, Shizuoka
  - Shizuoka, Shizuoka
  - Narutochō-mitsuishi, Tokushima
  - Tokushima, Tokushima
  - Edogawa-ku, Tokyo
  - Hachiōji, Tokyo
  - Higashikurume, Tokyo
  - Itabashi-ku, Tokyo
  - Meguro-ku, Tokyo
  - Ōta-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Tottori-shi, Tottori
  - Toyama, Toyama
  - Wakayama, Wakayama
  - Higashikawada, Yamagata
  - Shimonoseki, Yamaguchi
  - Shūnan, Yamaguchi

REFERENCES:
- [Result] Hori M, Matsumoto M, Tanahashi N, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iwamoto K, Tajiri M; J-ROCKET AF study investigators. Rivaroxaban vs. warfarin in Japanese patients with atrial fibrillation - the J-ROCKET AF study -. Circ J. 2012;76(9):2104-11. doi: 10.1253/circj.cj-12-0454. Epub 2012 Jun 5. PMID 22664783
- [Result] Chan MY, Lin M, Lucas J, Moseley A, Thompson JW, Cyr D, Ueda H, Kajikawa M, Ortel TL, Becker RC. Plasma proteomics of patients with non-valvular atrial fibrillation on chronic anti-coagulation with warfarin or a direct factor Xa inhibitor. Thromb Haemost. 2012 Dec;108(6):1180-91. doi: 10.1160/TH12-05-0310. Epub 2012 Oct 10. PMID 23052711
- [Result] Tanahashi N, Hori M, Matsumoto M, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iwamoto K, Tajiri M; J-ROCKET AF Study Investigators. Rivaroxaban versus warfarin in Japanese patients with nonvalvular atrial fibrillation for the secondary prevention of stroke: a subgroup analysis of J-ROCKET AF. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):1317-25. doi: 10.1016/j.jstrokecerebrovasdis.2012.12.010. Epub 2013 Jan 22. PMID 23352688
- [Result] Hori M, Matsumoto M, Tanahashi N, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iwamoto K, Tajiri M; J-ROCKET AF study investigators. Safety and efficacy of adjusted dose of rivaroxaban in Japanese patients with non-valvular atrial fibrillation: subanalysis of J-ROCKET AF for patients with moderate renal impairment. Circ J. 2013;77(3):632-8. doi: 10.1253/circj.cj-12-0899. Epub 2012 Dec 8. PMID 23229461
- [Result] Tanigawa T, Kaneko M, Hashizume K, Kajikawa M, Ueda H, Tajiri M, Paolini JF, Mueck W. Model-based dose selection for phase III rivaroxaban study in Japanese patients with non-valvular atrial fibrillation. Drug Metab Pharmacokinet. 2013;28(1):59-70. doi: 10.2133/dmpk.dmpk-12-rg-034. Epub 2012 Jul 17. PMID 22813718
- [Result] Kaneko M, Tanigawa T, Hashizume K, Kajikawa M, Tajiri M, Mueck W. Confirmation of model-based dose selection for a Japanese phase III study of rivaroxaban in non-valvular atrial fibrillation patients. Drug Metab Pharmacokinet. 2013;28(4):321-31. doi: 10.2133/dmpk.dmpk-12-rg-109. Epub 2013 Jan 22. PMID 23337693
- [Result] Matsumoto M, Hori M, Tanahashi N, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iekushi K, Yamanaka S, Tajiri M; J-ROCKET AF Study Investigators. Rivaroxaban versus warfarin in Japanese patients with non-valvular atrial fibrillation in relation to hypertension: a subgroup analysis of the J-ROCKET AF trial. Hypertens Res. 2014 May;37(5):457-62. doi: 10.1038/hr.2014.1. Epub 2014 Jan 30. PMID 24477179
- [Result] Uchiyama S, Hori M, Matsumoto M, Tanahashi N, Momomura S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iekushi K, Yamanaka S, Tajiri M; J-ROCKET AF Study Investigators. Net clinical benefit of rivaroxaban versus warfarin in Japanese patients with nonvalvular atrial fibrillation: a subgroup analysis of J-ROCKET AF. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):1142-7. doi: 10.1016/j.jstrokecerebrovasdis.2013.10.001. Epub 2013 Nov 1. PMID 24189454
- [Result] Hori M, Matsumoto M, Tanahashi N, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iekushi K, Yamanaka S, Tajiri M; J-ROCKET AF Study Investigators. Rivaroxaban versus warfarin in Japanese patients with nonvalvular atrial fibrillation in relation to the CHADS2 score: a subgroup analysis of the J-ROCKET AF trial. J Stroke Cerebrovasc Dis. 2014 Feb;23(2):379-83. doi: 10.1016/j.jstrokecerebrovasdis.2013.07.021. Epub 2013 Aug 15. PMID 23954611
- [Result] Hori M, Kajikawa M. The J-ROCKET AF Study: a matter of ethnicity or a matter of weight? Reply. Circ J. 2013;77(10):2637. doi: 10.1253/circj.cj-13-0879. Epub 2013 Aug 1. No abstract available. PMID 23903065
- [Result] Hori M, Matsumoto M, Tanahashi N, Momomura S, Uchiyama S, Goto S, Izumi T, Koretsune Y, Kajikawa M, Kato M, Ueda H, Iekushi K, Yamanaka S, Tajiri M; J-ROCKET AF Study Investigators. Rivaroxaban vs. warfarin in Japanese patients with non-valvular atrial fibrillation in relation to age. Circ J. 2014;78(6):1349-56. doi: 10.1253/circj.cj-13-1324. Epub 2014 Apr 7. PMID 24705469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 08 Jun 2007, and the last participant completed the study on 19 Jan 2010. The study was conducted at 167 centers in Japan. 164 study centers enrolled at least 1 participant.
Pre-assignment Details: In total, 1439 participants were screened for study eligibility; 159 participants were screening failures and were not randomized. Therefore, 1280 participants (640 in each group) were randomized.
Period: Double-blind (DB) Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Started | 640 | 640
Started Treatment | 639 (Safety population) | 639 (Safety population)
Completed | 480 | 468
Not Completed | 160 | 172
Not completed — Adverse Event | 73 | 70
Not completed — Withdrawal by Subject | 26 | 35
Not completed — Death | 8 | 3
Not completed — Physician Decision | 4 | 13
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 9 | 9
Not completed — Clinical Endpoint Reached | 18 | 28
Not completed — Non-compliant with Study Medication | 3 | 1
Not completed — Protocol Driven Decision Point | 12 | 8
Not completed — Site Closed by Investigator | 1 | 2
Not completed — Site Closed by Sponsor | 1 | 1
Not completed — Drop out before Treatment Start | 1 | 1
Period: Follow-up (FU) Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Started | 639 (All treated participants were to enter FU period, whether or not they completed the DB period) | 639 (All treated participants were to enter FU period, whether or not they completed the DB period)
Entered FU and Valid for Safety | 628 (Safety population) | 630 (Safety population)
Completed | 610 | 616
Not Completed | 29 | 23
Not completed — Adverse Event | 1 | 1
Not completed — Death | 13 | 12
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Clinical Endpoint Reached | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin | Total
Number analyzed (Participants) | 640 | 640 | 1280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (8.3) | 71.2 (7.9) | 71.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 140 | 250
  Male | 530 | 500 | 1030
CL(CR) [creatinine clearance] [Number; unit: Participants]
  <50 mL/min | 141 | 143 | 284
  50 to <80 mL/min | 329 | 329 | 658
  ≥80 mL/min | 170 | 168 | 338

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of the Composite Endpoint of Adjudicated Major Bleeding or Adjudicated Non-major Clinically Relevant Bleeding
Description: Major bleeding: clinically overt bleeding (COB) associated with a fall in hemoglobin ≥2 g/dL, leading to transfusion ≥2 units of packed red blood cells or whole blood, occurring in a critical site or contributing to death. Non-major clinically relevant bleeding: COB that does not meet the definition of major bleeding, but requires medical intervention or unscheduled contact with the physician, (temporary) discontinuation of the study treatment, discomfort to the subject such as pain, or impairment of activities of daily life.
Time Frame: Up to 2 days after the last dose
Population: The safety analysis population consisted of randomized participants who took at least one dose of study treatment (639 in each treatment group).
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 639 | 639
Events per 100 patient-years | 18.04 | 16.42
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 2.0; p = 0.025, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.87 to 1.42]

2. Secondary Outcome: Event Rate of the Composite Endpoint of Adjudicated Stroke and Non-central Nervous System (CNS) Systemic Embolism
Description: This is the principal efficacy endpoint. Stroke included hemorrhagic, ischemic infarction and unknown. Arterial emboli in the following areas were "non-CNS systemic embolism": peripheral arterial in the upper and lower extremities, renal, mesenteric, splenic, hepatic, ocular/retinal and others. Pulmonary embolism or myocardial infarction was excluded.
Time Frame: Up to 2 days after the last dose
Population: The per-protocol analysis population consisted of randomized participants excluding those who had specific pre-defined major protocol deviations (637 in each treatment group).
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 1.26 | 2.61
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.24 to 1.00]

3. Secondary Outcome: Event Rate of the Composite Endpoint of Adjudicated Stroke, Non-CNS Systemic Embolism, and Vascular Death
Description: Stroke included hemorrhagic, ischemic infarction and unknown. Arterial emboli in the following areas were "non-CNS systemic embolism": peripheral arterial in the upper and lower extremities, renal, mesenteric, splenic, hepatic, ocular/retinal and others. Pulmonary embolism or myocardial infarction was excluded. Any death that was not clearly non-vascular.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 1.83 | 2.85
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.34 to 1.22]

4. Secondary Outcome: Event Rate of the Composite Endpoint of Adjudicated Stroke, Non-CNS Systemic Embolism, Myocardial Infarction, and Vascular Death
Description: Stroke included hemorrhagic, ischemic infarction and unknown. Arterial emboli in the following areas were "non-CNS systemic embolism": peripheral arterial in the upper and lower extremities, renal, mesenteric, splenic, hepatic, ocular/retinal and others. Pulmonary embolism or myocardial infarction was excluded. Myocardial infarction: assessed based on either cardiac biomarkers, new abnormal Q waves appeared on electrocardiogram for ≥2 leads, or autopsy confirmation. Any death that was not clearly non-vascular.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 2.18 | 2.97
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.41 to 1.34]

5. Secondary Outcome: Event Rate of Stroke
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Stroke included hemorrhagic (Stroke with local collections of intraparenchymal blood. Subarachnoid hemorrhage, subdural hemorrhage, and epidural hemorrhage were excluded.), ischemic infarction (Stroke without focal collection of intracranial blood) and unknown (No imaging data and anatomic findings were available.).
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 1.15 | 2.49
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.22 to 0.98]

6. Secondary Outcome: Event Rate of Non-CNS Systemic Embolism
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Non-CNS systemic embolism was abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms (such as trauma, atherosclerosis, and instrumentation). Arterial emboli in the following areas were "non-CNS systemic embolism": peripheral arterial in the upper and lower extremities, renal, mesenteric, splenic, hepatic, ocular/retinal and others. Pulmonary embolism or myocardial infarction was excluded from this category.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 0.11 | 0.12
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.06 to 15.85]

7. Secondary Outcome: Event Rate of Myocardial Infarction
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Myocardial infarction was assessed based on either cardiac bio-markers (troponin I, troponin T, or creatine kinase-muscle and brain subunit isozyme), new abnormal Q waves appeared on ECG for 2 or more leads, or autopsy confirmation.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 0.34 | 0.12
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 2.93, 95% CI 2-sided [0.30 to 28.16]

8. Secondary Outcome: Event Rate of Vascular Death
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Any death that was not clearly non-vascular (e.g., deaths due to spontaneous bleeding, myocardial infarction, stroke, cardiac failure, and arrhythmia)
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 0.69 | 0.24
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 2.97, 95% CI 2-sided [0.60 to 14.70]

9. Secondary Outcome: Event Rate of Stroke With Serious Residual Disability
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. A stroke was considered disabling if the participant's modified Rankin score was between 3 and 5, inclusive.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 0.57 | 1.19
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.16 to 1.40]

10. Secondary Outcome: Event Rate of All-cause Death
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. All-cause death included vascular death and non-vascular death.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 2
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 637 | 637
Events per 100 patient-years | 0.80 | 0.59
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.43 to 4.31]

11. Secondary Outcome: Event Rate of Adjudicated Major Bleeding
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Major bleeding was clinically overt bleeding associated with a fall in hemoglobin of 2 g/dL or higher, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 1
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 639 | 639
Events per 100 patient-years | 3.00 | 3.59
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.50 to 1.43]

12. Secondary Outcome: Event Rate Adjudicated Non-major Clinically Relevant Bleeding
Description: All events were adjudicated and confirmed by a central independent committee blinded to treatment. Non-major clinically relevant bleeding was clinically overt bleeding that does not meet the definition of major bleeding, but requires medical intervention or unscheduled contact with the physician, (temporary) discontinuation of the study treatment, discomfort to the subject such as pain, or impairment of activities of daily life.
Time Frame: Up to 2 days after the last dose
Population: as for outcome 1
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin
Number analyzed (Participants) | 639 | 639
Events per 100 patient-years | 15.42 | 12.99
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin; Test type: Superiority or Other; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.92 to 1.56]

ADVERSE EVENTS:
Time Frame: Reporting Group (RG) 1 + 2: Safety data collected start with the first dose of study drug up to 2 days after the last dose; Reporting Group (RG) 3 + 4: Safety data collected from last dose plus 2 days to end of trial.
Description: RG3: During follow-up period, participants could be transitioned from study drug to an open-label warfarin or other appropriate therapy.
Groups:
- RG1: Rivaroxaban Double-blind (DB) Period: Participants orally administered a rivaroxaban 15 mg tablet (a 10 mg tablet for participants with creatinine clearance of 30 to 49 mL/min, inclusive, at screening) and a warfarin placebo tablet once daily (OD) during the double-blind treatment period. Safety data collected start with the first dose of study drug up to 2 days after the last dose
- RG2: Warfarin DB Period: Participants orally administered a warfarin potassium tablet and a rivaroxaban placebo tablet OD during the double-blind treatment period. Safety data collected start with the first dose of study drug up to 2 days after the last dose
- RG3: Rivaroxaban Follow-up (FU) Period: Participants orally administered a rivaroxaban 15 mg tablet (a 10 mg tablet for participants with creatinine clearance of 30 to 49 mL/min, inclusive, at screening) and a warfarin placebo tablet once daily (OD) during the double-blind treatment period. Safety data collected from last dose plus 2 days to end of trial
- RG4: Warfarin FU Period: Participants orally administered a warfarin potassium tablet and a rivaroxaban placebo tablet OD during the double-blind treatment period. Safety data collected from last dose plus 2 days to end of trial
Arm/Group | RG1: Rivaroxaban Double-blind (DB) Period | RG2: Warfarin DB Period | RG3: Rivaroxaban Follow-up (FU) Period | RG4: Warfarin FU Period
Serious Adverse Events (participants affected / at risk) | 151/639 | 155/639 | 50/628 | 37/630
Other Adverse Events (participants affected / at risk) | 474/639 | 470/639 | 73/628 | 61/630
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RG1: Rivaroxaban Double-blind (DB) Period (N=639) | RG2: Warfarin DB Period (N=639) | RG3: Rivaroxaban Follow-up (FU) Period (N=628) | RG4: Warfarin FU Period (N=630)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 12 (12) | 11 (18) | 3 (3) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Auditory meatus external erosion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 9 (10) | 7 (8) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 5 (5) | 9 (12) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 14 (15) | 10 (11) | 3 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (6) | 2 (2) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cholinergic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 9 (9) | 18 (18) | 10 (12) | 4 (4)
Postresuscitation encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosomatic disease (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal embolism (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (5) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis obliterans (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RG1: Rivaroxaban Double-blind (DB) Period (N=639) | RG2: Warfarin DB Period (N=639) | RG3: Rivaroxaban Follow-up (FU) Period (N=628) | RG4: Warfarin FU Period (N=630)
Cardiac failure (Cardiac disorders) | 36 (39) | 29 (35) | 5 (6) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 26 (32) | 42 (57) | 9 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 38 (46) | 32 (40) | 12 (12) | 8 (8)
Dental caries (Gastrointestinal disorders) | 28 (32) | 34 (35) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 57 (71) | 40 (47) | 3 (3) | 6 (6)
Gingival bleeding (Gastrointestinal disorders) | 54 (72) | 31 (38) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 206 (378) | 232 (412) | 16 (16) | 15 (16)
Contusion (Injury, poisoning and procedural complications) | 58 (82) | 56 (80) | 4 (4) | 4 (4)
Wound haemorrhage (Injury, poisoning and procedural complications) | 33 (38) | 27 (31) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 43 (48) | 31 (34) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (57) | 56 (60) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 24 (29) | 39 (43) | 6 (6) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 102 (203) | 59 (86) | 6 (8) | 8 (8)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 55 (76) | 74 (102) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 37 (50) | 43 (49) | 2 (2) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 67 (147) | 79 (175) | 9 (9) | 6 (7)
Hypertension (Vascular disorders) | 24 (25) | 32 (36) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less